CLINICAL TRIAL: NCT05180812
Title: Safety and Feasibility of Upper Extremity ExoNET Support Post Stroke
Brief Title: Safety and Feasibility of ExoNET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Lanphier Patton, Co-Director, Robotics Laboratory, Arms and Hands Lab, Shirley Ryan AbilityLab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00216062
Record Dates: First submitted 2021-12-05; First posted 2022-01-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Cerebral Vascular Accident
Keywords: Upper Extremity; Rehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: Gravity Compensation (Experimental): The participants will be wearing the ExoNet device tuned to gravity support.
  Interventions: Device: ExoNet Tuned to Gravity Support
- Control Group: No Gravity Compensation (Sham Comparator): The participants will be wearing the ExoNet device, but it will not be tuned to gravity support.
  Interventions: Device: ExoNet Tuned to Gravity Support

INTERVENTIONS:
Device: ExoNet Tuned to Gravity Support — This study's primary goal is to test the safety, feasibility, and efficacy of the ExoNET device developed in the Robotics Lab at the Shirley Ryan AbilityLab. We want to observe if individuals using the ExoNET tuned to gravity support will notice a reduction in bicep muscle activity, leading to an improvement in functional outcome measures in stroke patients.

SUMMARY:
The purpose of this study is to evaluate the safety, feasibility, and preliminary efficacy of the ExoNET passive robotic device. It will provide upper-extremity gravity compensation for therapeutic movement retraining in the chronic post stroke patient population.

DETAILED DESCRIPTION:
The ExoNET, a passive robotic solution that provides a soft, biomimetic, and elastic alternative to robotics that embodies intelligence within the mechanical design. Several groups have been exploring performance enhancement using springs with custom-tuned parameters via optimization. Here, it is possible to have a simple reconfigurable system that can not only assist performance, but can also make training easier, faster, and more complete. This contribution has the potential to be clinically significant for rehabilitating neurologically impaired individuals because this proposal will investigate how motor learning can be facilitated through novel assistive technology.

The primary objective of this study is to evaluate the safety, feasibility and efficacy using the ExoNET. Specifically, investigators want to see if the ExoNET tuned to gravity support will lead to a reduction in bicep muscle activity and an increase in range of motion. To accomplish this aim, we plan to have participants perform reaching, arm elevation and flexion task exercises wearing the ExoNET. To achieve these goals, we will use a wearable activity tracker (MiGo), to detect the number of activities performed, a wearable surface EMG system (Delsys) on the bicep muscles and a markerless system called the Kinect (version 2) to collect distribution of motion.

Investigators hypothesize that individuals with post-stroke arm movement deficits treated with ExoNET gravity compensation will improve their ARAT measures more than controls receiving a sham treatment. Secondarily, treated subjects will improve in other clinical metrics and will make more movements than controls.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrhagic stroke (8 months post stroke)
2. Available medical records and radiographic information about lesion locations
3. Hemiparesis
4. Some degree of both shoulder and elbow movement capability
5. A "moderate" impairment (Fugl-Meyer score between 15-50)

Exclusion Criteria:

1. Individuals under the age of 18
2. Bilateral paresis
3. Shoulder pain and/or articular rigidity on the upper limb joint
4. Spasticity (Modified Ashworth Scale of 2)
5. Botox injection to the affected upper extremity within the previous 4 months
6. Aphasia, cognitive impairment, or affective dysfunction that would influence the ability to perform the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2026-07-12 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test | Tested at week 1 (baseline evaluations), week 4 (post evaluations), and week 9 (follow-up evaluations)
  observational measure used to assess change in upper extremity performance in individuals with a damaged nervous system

SECONDARY OUTCOMES:
Fugl-Meyer | Tested at week 1 (baseline evaluations), week 4 (post evaluations), and week 9 (follow-up evaluations)
  observational measure used to measure change in upper extremity impairment in individuals with a damaged nervous system
Wolf Motor Function Test | Tested at week 1 (baseline evaluations), week 4 (post evaluations), and week 9 (follow-up evaluations)
  Quantitative measure of change of upper extremity motor ability
Box and Blocks | Tested at week 1 (baseline evaluations), week 4 (post evaluations), and week 9 (follow-up evaluations)
  Measures change in unilateral gross motor dexterity

OTHER OUTCOMES:
Electromyography using Delsys | Treatment phases (week 2 and week 3)
  Delsys sensors will be used to measure change in biceps activity
Kinect | Treatment phases (week 2 and week 3)
  markerless system to collect changes of distribution of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celian C, Ryali P, Wilson V, Srivatsa A, Patton JL. A Wearable Anti-Gravity Supplement to Therapy Does Not Improve Arm Function in Chronic Stroke: A Randomized Pilot Trial. Neurorehabil Neural Repair. 2025 Sep;39(9):728-741. doi: 10.1177/15459683251338792. Epub 2025 Jun 19. PMID 40537460